CLINICAL TRIAL: NCT00153465
Title: University of Oklahoma Health Sciences Center Parenting Program Attrition and Compliance Efficacy Trial
Brief Title: University of Oklahoma Parenting Program Attrition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CDC-NCIPC-3899; R49/CCR622338-04
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Child Abuse
Keywords: Parent training; Child maltreatment; Motivation; Program attrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Motivational intervention, parent training

SUMMARY:
The study will examine the extent to which a group motivational intervention (ME) impacts retention, treatment compliance, and long-term outcomes in families with a history of, or high risk for, child maltreatment.

DETAILED DESCRIPTION:
The field of child abuse prevention faces not only the challenge of developing and disseminating effective treatments, but the problem of high attrition rates and treatment noncompliance. This study will compare the effects of a motivational intervention with a "services as usual" orientation group on program retention, treatment compliance, and long-term outcomes in families with histories of child maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* Families referred to service agency for child maltreatment prevention services
* Families with children between 2-1/2 and 12 years of age

Exclusion Criteria:

* Parents with cognitive, psychiatric, or social conditions that would limit their ability to provide voluntary consent or benefit from the intervention
* Parents who have sexually abused their children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2004-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Incidents of child maltreatment 1-3 years post-treatment

SECONDARY OUTCOMES:
Parenting behaviors, attitudes, and functioning assessed during and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Chaffin, Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States